CLINICAL TRIAL: NCT04667416
Title: A Prospective, Multicenter, Randomized, Controlled Clinical Investigation of PalinGen® Flow Amniotic Tissue Allograft to Assess Safety, Tolerability, and Preliminary Efficacy for the Treatment of Chronic Lower Extremity Cutaneous Ulcers Compared to Standard of Care
Brief Title: Safety and Preliminary Efficacy of PalinGen Flow Amniotic Tissue Allograft in Chronic Ulcers of the Lower Extremities
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Amnio Technology, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PGF-201
Record Dates: First submitted 2020-12-08; First posted 2020-12-14 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Chronic Ulcer of Lower Extremity
Keywords: Diabetic ulcer; Venous stasis ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SOC) (No Intervention): Participants will receive SOC for chronic ulcers of the lower extremities.
- PalinGen Flow Treatment plus SOC (Experimental): Participants will receive wound size-dependent dose of PalinGen Flow liquid human amniotic tissue allograft by subcutaneous injection in addition to SOC.
  Interventions: Biological: PalinGen Flow Amniotic Tissue Allograft

INTERVENTIONS:
Biological: PalinGen Flow Amniotic Tissue Allograft — Participants will receive wound size-dependent dose of PalinGen Flow liquid human amniotic tissue allograft by subcutaneous injection in addition to SOC.
  Arms: PalinGen Flow Treatment plus SOC

SUMMARY:
The purpose of this study is to assess the safety and preliminary efficacy of PalinGen® Flow for the treatment of chronic ulcers of the lower legs and feet.

ELIGIBILITY:
Inclusion Criteria:

* Able to read, understand and sign the informed consent form (ICF)
* Available and willing to complete all study assessments
* At least 12 weeks post lower extremity revascularization procedure, if one has been performed
* Have chronic ulcer(s) of the lower extremities with the following characteristics:

  * Of diabetic or vascular etiology
  * Duration of ≥4 weeks, unresponsive to SOC
  * ≤20 cm2 in area
  * Extend through the full thickness of the skin but not down to muscle, tendon, or bone
* For subjects with VLU:

  * Ulcer area is ≥1.5 cm2 and ≤20 cm2 and with a clean, granulating base with minimal adherent slough
  * Ulcer location is at or above the ankle (malleolus) and below the knee
  * Ulcer location is appropriate for use of compression therapy treatment
* For subjects with DFU:

  * Ulcer area is ≥1.5 cm2 and ≤ 20 cm2 and is amenable to off-loading
  * Subject has diabetes mellitus (Type 1 or Type 2), requiring insulin or oral/injectable medications to control blood glucose levels
  * Glycosylated hemoglobin (HbA1c) level at screening is <12%
* Adequate circulation to the affected lower extremities
* Total serum bilirubin, alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST), hemoglobin, WBC, and PLT count all within limits specified in study protocol
* No renal impairment or mild renal impairment, defined as creatinine clearance ≥50 mL/min (by Cockroft-Gault estimation)
* Male subjects and female subjects of childbearing potential must use acceptable methods of contraception

Exclusion Criteria:

* Clinical evidence of ongoing infection and/or receipt of IV, oral, or topical antimicrobials at the Baseline Visit
* Wheelchair bound or bed-ridden (ambulatory with assistance is acceptable)
* Ulceration at the site of amputation
* Undergoing renal dialysis
* Known or suspected malignancy in the target ulcer, or a history of cancer in the preceding 5 years (other than carcinoma in situ of the cervix or adequately treated non-melanoma skin cancer)
* Documented history of osteomyelitis at the target ulcer location within 6 months of screening
* Current treatment or anticipated need for treatment over the course of the study with:

  * Immunosuppressants (including topical or systemic corticosteroids or glucocorticoids)
  * Cytotoxic chemotherapy
  * Growth hormone
  * Oral or systemic antifungal or antituberculosis treatment
* History of radiation at the ulcer site
* New York Heart Association Class III or IV congestive heart failure or uncontrolled cardiac dysrhythmia
* Diagnosis of autoimmune disease(s) (rheumatoid arthritis, lupus, psoriasis, Sjogren's syndrome) or arthritis requiring corticosteroid treatment
* Target ulcer(s) previously treated with negative pressure, hyperbaric oxygen, or tissue engineered materials (eg, Apligraf®, EpiFix® or Dermagraft®) or other scaffold materials (eg, Oasis, Matristem) within 4 weeks prior to Screening Visit
* Target ulcer(s) anticipated to require negative pressure wound therapy or hyperbaric oxygen at any time during the study
* Subjects with VLU who have:

  * Deep vein thrombosis diagnosed within 4 weeks prior to Screening Visit
  * Refusal or inability to tolerate compression therapy
* Subjects with DFU who have:

  * Active Charcot foot (stable chronic Charcot foot is not exclusionary)
  * Ulcers on toes 2, 3, 4, and/or 5 only (ulcer on plantar surface of the great toe only is not exclusionary)
* Pregnant or breast feeding
* Allergic to DMSO
* Healing of target ulcer is observed to be ≥35% at the end of the Run-in Period (between Screening and Baseline Visits)
* Presence of any condition(s) which compromises the subject's ability to complete this study, including subjects with a known history of poor adherence to medical treatment
* Subjects who, in the opinion of the Investigator, are not able to comply with study requirements
* Treatment with an investigational drug(s) or device(s) within the 4 weeks preceding Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants in the PalinGen Flow plus SOC group versus SOC alone with treatment-emergent adverse events (TEAEs) | All adverse events (AEs) and serious adverse events (SAEs) will be recorded from the time of signing of the informed consent form through Week 64.
  Treatment-emergent adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) and graded per the CTCAE Version 5.0.
Proportion of participants in the PalinGen Flow plus SOC group versus SOC alone who achieve complete ulcer closure by Week 12. | BWAT assessment and wound imaging will be performed at each study visit through end of treatment (Week 12)
  Complete wound closure will be assessed by the Bates-Jensen Wound Assessment Tool (BWAT) and a photographic imaging and measurement device.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Caporusso, D.P.M., Principal Investigator — Futuro Clinical Trials
Locations (7):
- United States (7):
  - Center for Clinical Research, Carmichael, California
  - Center for Clinical Research, Castro Valley, California
  - Limb Preservation Platform, Fresno, California
  - Center for Clinical Research, San Francisco, California
  - ILD Research Center, Vista, California
  - Acclaim Bone & Joint Institute and Plastic Surgery, Fort Worth, Texas
  - Futuro Clinical Trials, McAllen, Texas